CLINICAL TRIAL: NCT03181789
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of pDNA Vaccines Expressing HIV M Group p24^Gag Conserved Elements and/or p55^Gag, Administered With IL-12 pDNA, in Healthy, HIV-Uninfected Adult Participants
Brief Title: Safety and Immunogenicity of pDNA Vaccines Expressing HIV M Group p24^Gag Conserved Elements and/or p55^Gag, Administered With IL-12 pDNA
Acronym: HVTN119
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 119; 12061 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: HIV Infections
Keywords: HIV vaccine; DNA vaccine; IL-12; Electroporation; p24; Gag; Adjuvant; Healthy
MeSH Terms: conditions — HIV Infections | interventions — Electroporation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Group 1 (Treatment): p24CE1/2 pDNA + p55^gag pDNA + IL-12 pDNA (Experimental): Participants will receive the p24CE1/2 pDNA vaccine and the IL-12 pDNA adjuvant at Day 0 and Month 1. They will receive the p24CE1/2 pDNA vaccine plus the p55^gag pDNA vaccine and the IL-12 pDNA adjuvant at Months 3 and 6.
  Interventions: Biological: p24CE1/2 pDNA Vaccine; Biological: p55^gag pDNA Vaccine; Biological: IL-12 pDNA Adjuvant; Device: Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device
- Group 1 (Control): Placebo (Placebo Comparator): Participants will receive placebo at Day 0 and Months 1, 3, and 6.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device
- Group 2 (Treatment): p55^gag pDNA + IL-12 pDNA (Experimental): Participants will receive the p55^gag pDNA vaccine and the IL-12 pDNA adjuvant at Day 0 and Months 1, 3, and 6.
  Interventions: Biological: p55^gag pDNA Vaccine; Biological: IL-12 pDNA Adjuvant; Device: Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device
- Group 2 (Control): Placebo (Placebo Comparator): Participants will receive placebo at Day 0 and Months 1, 3, and 6.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device

INTERVENTIONS:
Biological: p24CE1/2 pDNA Vaccine — Administered bilaterally using the Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device
  Other Names: p24CE1/2
  Arms: Group 1 (Treatment): p24CE1/2 pDNA + p55^gag pDNA + IL-12 pDNA
Biological: p55^gag pDNA Vaccine — Administered bilaterally using the TDS-IM EP device
  Other Names: p55^gag
  Arms: Group 1 (Treatment): p24CE1/2 pDNA + p55^gag pDNA + IL-12 pDNA; Group 2 (Treatment): p55^gag pDNA + IL-12 pDNA
Biological: IL-12 pDNA Adjuvant — Administered bilaterally using the TDS-IM EP device
  Other Names: GENEVAX® IL-12 DNA Plasmid
  Arms: Group 1 (Treatment): p24CE1/2 pDNA + p55^gag pDNA + IL-12 pDNA; Group 2 (Treatment): p55^gag pDNA + IL-12 pDNA
Biological: Placebo — Administered bilaterally using the TDS-IM EP device
  Arms: Group 1 (Control): Placebo; Group 2 (Control): Placebo
Device: Ichor Medical Systems Intramuscular TriGrid Delivery System (TDS-IM) electroporation (EP) device — The TDS-IM EP device will be used to administer study product(s).
  Other Names: TDS-IM EP device

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of two HIV-1 pDNA vaccines: p24CE1/2 pDNA and p55^gag pDNA administered with IL-12 pDNA adjuvant, given by intramuscular (IM) injection with electroporation (EP), in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity of two HIV-1 pDNA vaccines: p24CE1/2 pDNA and p55^gag pDNA administered with IL-12 pDNA adjuvant, given by intramuscular (IM) injection with electroporation (EP), in healthy, HIV-uninfected adults.

Participants will be randomly assigned to one of four groups: Group 1 Treatment, Group 1 Control, Group 2 Treatment, or Group 2 Control.

Participants in Group 1 Treatment will receive p24CE1/2 pDNA and IL-12 pDNA at Day 0 and Month 1, then p24CE1/2 pDNA plus p55^gag pDNA and IL-12 pDNA at Months 3 and 6. Participants in Group 1 Control will receive placebo (sodium chloride for injection) at Day 0 and Months 1, 3, and 6.

Participants in Group 2 Treatment will receive p55^gag pDNA and IL-12 pDNA at Day 0 and Months 1, 3, and 6. Participants in Group 2 Control will receive placebo (sodium chloride for injection) at Day 0 and Months 1, 3, and 6.

Study visits will occur at Day 0, Week 2, and Months 1, 1.25, 1.5, 3, 3.5, 6, 6.25, 6.5, 9, and 12. Visits may include physical examinations and clinical assessments, blood and urine collection, optional stool collection, HIV testing, risk reduction counseling, and interviews/questionnaires. At Month 18, study staff will contact participants for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol visit (excludes annual health contact visit)
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatine phosphokinase (CPK) less than or equal to 2.0 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: U.S. volunteers must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin

Reproductive Status

* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit.
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.

Exclusion Criteria:

General

* Allergy to amide-type local anesthetics (bupivacaine [Marcaine], lidocaine [Xylocaine], mepivacaine [Polocaine/Carbocaine], etidocaine [Duranest], prilocaine [Citanest, EMLA® cream])
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the study
* Pregnant or breastfeeding
* Active duty and reserve U.S. military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 119 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial.

Immune System

* Immunosuppressive medications received within 168 days before first vaccination.
* Serious adverse reactions to vaccines or to vaccine components
* Autoimmune disease
* Immunodeficiency

Clinically significant medical conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy
* Seizure disorder
* Asplenia
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Presence of implanted electronic medical device (e.g., cochlear implant, pacemaker, implantable cardioverter defibrillator)
* Presence of surgical or traumatic metal implant at the intended site of administration (including the deltoid muscles and/or overlying skin)
* Sinus bradycardia (defined as less than 50 beats per minute (bpm) on exam) or a history of cardiac arrhythmia: e.g., supraventricular tachycardia, atrial fibrillation, or frequent ectopy. NOTE: Sinus arrhythmia is not excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kalams, Study Chair — Vanderbilt University; Hyman Scott, Study Chair — Bridge HIV, SFDPH
Locations (3):
- United States (3):
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Case Clinical Research Site, Cleveland, Ohio

REFERENCES:
- [Derived] Kalams SA, Felber BK, Mullins JI, Scott HM, Allen MA, De Rosa SC, Heptinstall J, Tomaras GD, Hu J, DeCamp AC, Rosati M, Bear J, Pensiero MN, Eldridge J, Egan MA, Hannaman D, McElrath MJ, Pavlakis GN; HIV Vaccine Trials Network 119(HVTN 119) Study Team. Focusing HIV-1 Gag T cell responses to highly conserved regions by DNA vaccination in HVTN 119. JCI Insight. 2024 Aug 1;9(18):e180819. doi: 10.1172/jci.insight.180819. PMID 39088271

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: P24CE1/2(CE/CE) + gag vaccines
- Group 2: Vaccine: P55gag (gag/gag) vaccines
- Group 3: Control 1; Group 4: Control 2: Placebo: Sodium Chloride, USP 0.9%
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Started | 25 | 25 | 3 | 3
Safety Population | 25 | 25 | 3 | 3
Completed | 18 | 22 | 2 | 3
Not Completed | 7 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 7 | 1 | 0 | 0
Not completed — Participant unable to adhere to visit | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2 | Total
Number analyzed (Participants) | 25 | 25 | 3 | 3 | 56
Age, Continuous [Median (Full Range); unit: years] | 29 [20 to 50] | 31 [18 to 47] | 24 [21 to 43] | 30 [23 to 35] | 29 [18 to 50]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 | 0 | 0 | 0 | 0 | 0
  18 - 20 | 1 | 1 | 0 | 0 | 2
  21 - 30 | 13 | 11 | 2 | 2 | 28
  31 - 40 | 3 | 9 | 0 | 1 | 13
  41 - 50 | 8 | 4 | 1 | 0 | 13
  Over 50 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 3 | 3 | 33
  Male | 13 | 10 | 0 | 0 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 0 | 5
  Not Hispanic or Latino | 24 | 22 | 2 | 3 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 4 | 6 | 0 | 0 | 10
  White | 16 | 11 | 3 | 3 | 33
  More than one race | 2 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 3 | 3 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. The maximum grade observed for each symptom ove
Time Frame: Measured through Month 0, 1, 3, 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  Pain: None | 4 | 1 | 0 | 0
  Pain: Mild | 13 | 21 | 2 | 3
  Pain: Moderate | 8 | 3 | 1 | 0
  Pain: Severe | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 0 | 0 | 0 | 0
  Tenderness: Mild | 17 | 18 | 1 | 2
  Tenderness: Moderate | 8 | 7 | 2 | 1
  Tenderness: Severe | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Mild | 15 | 18 | 1 | 2
  Pain and/or Tenderness: Moderate | 10 | 7 | 2 | 1
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through Month 0, 1, 3, 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  Erythema/Redness: None | 23 | 21 | 2 | 2
  Erythema/Redness: Mild | 2 | 3 | 1 | 1
  Erythema/Redness: Moderate | 0 | 1 | 0 | 0
  Erythema/Redness: Severe | 0 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Induration/Swelling: None | 23 | 22 | 3 | 3
  Induration/Swelling: Mild | 1 | 2 | 0 | 0
  Induration/Swelling: Moderate | 1 | 1 | 0 | 0
  Induration/Swelling: Severe | 0 | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 22 | 20 | 2 | 2
  Erythema and/or Induration: Mild | 2 | 4 | 1 | 1
  Erythema and/or Induration: Moderate | 1 | 1 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month 0, 1, 3, 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  Malaise and/or fatigue: None | 10 | 6 | 2 | 0
  Malaise and/or fatigue: Mild | 11 | 14 | 1 | 1
  Malaise and/or fatigue: Moderate | 3 | 4 | 0 | 2
  Malaise and/or fatigue: Severe | 1 | 1 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 13 | 15 | 0 | 0
  Myalgia: Mild | 9 | 8 | 3 | 2
  Myalgia: Moderate | 3 | 1 | 0 | 1
  Myalgia: Severe | 0 | 1 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 14 | 11 | 2 | 1
  Headache: Mild | 9 | 6 | 1 | 1
  Headache: Moderate | 2 | 7 | 0 | 1
  Headache: Severe | 0 | 1 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 18 | 18 | 3 | 2
  Nausea: Mild | 6 | 5 | 0 | 1
  Nausea: Moderate | 1 | 1 | 0 | 0
  Nausea: Severe | 0 | 1 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 25 | 24 | 3 | 3
  Vomiting: Mild | 0 | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 1 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 24 | 22 | 3 | 1
  Chills: Mild | 1 | 1 | 0 | 0
  Chills: Moderate | 0 | 1 | 0 | 2
  Chills: Severe | 0 | 1 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 19 | 21 | 2 | 1
  Arthralgia: Mild | 5 | 2 | 1 | 1
  Arthralgia: Moderate | 1 | 1 | 0 | 1
  Arthralgia: Severe | 0 | 1 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 4 | 3 | 0 | 0
  Max. Systemic Symptoms: Mild | 14 | 12 | 3 | 1
  Max. Systemic Symptoms: Moderate | 6 | 9 | 0 | 2
  Max. Systemic Symptoms: Severe | 1 | 1 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Temperature: None | 23 | 25 | 3 | 3
  Temperature: Mild | 2 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alkaline Phosphate (ALP), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Creatine Phosphokinase (CPK) in U/L
Description: For each local laboratory measure-alkaline phosphate (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatine phosphokinase (CPK) in U/L, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, Days 14, 42, 98, 182 and 273
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
U/L
  ALT (SGPT) (U/L)- Screening | 17 [12 to 23] | 16 [13 to 23] | 12 [9 to 15] | 16 [13 to 17]
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  ALT (SGPT) (U/L)-Day 14 | 14.5 [11 to 23] | 16.5 [11 to 21] | 9 [9 to 9] | 12 [10 to 15]
  ALT (SGPT) (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  ALT (SGPT) (U/L)-Day 42 | 14.5 [10.5 to 23] | 15 [12 to 22] | 12 [11 to 13] | 17 [11 to 38]
  ALT (SGPT) (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  ALT (SGPT) (U/L)-Day 98 | 15 [11 to 28] | 13 [11 to 22] | 11 [11 to 20] | 16 [14 to 20]
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  ALT (SGPT) (U/L)-Day 182 | 16 [13 to 21] | 17 [13 to 21] | 13 [12 to 17] | 13.5 [10 to 17]
  ALT (SGPT) (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  ALT (SGPT) (U/L)-Day 273 | 16 [13 to 22] | 15.5 [12 to 25.5] | 11 [11 to 11] | 12 [12 to 13]
  AST (U/L)- Screening | 17 [15 to 21] | 17 [15 to 22] | 18 [14 to 20] | 15 [12 to 29]
  AST (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  AST (U/L)-Day 14 | 16 [15 to 19.5] | 17 [15 to 19] | 13.5 [13 to 14] | 13 [13 to 16]
  AST (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  AST (U/L)-Day 42 | 16 [14 to 20] | 16 [15 to 20] | 14 [14 to 19] | 24 [13 to 62]
  AST (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  AST (U/L)-Day 98 | 17 [15 to 21] | 16 [15 to 19] | 15 [12 to 21] | 18 [16 to 22]
  AST (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  AST (U/L)-Day 182 | 18 [15 to 21] | 20 [15 to 24] | 17 [17 to 20] | 18 [15 to 21]
  AST (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 2
  AST (U/L)-Day 273 | 16 [15 to 21] | 18 [15.5 to 23] | 15.5 [15 to 16] | 15 [15 to 15]
  Alkaline Phosphatase (U/L)- Screening | 61 [48 to 72] | 61 [52 to 70] | 52 [51 to 55] | 54 [43 to 62]
  Alkaline Phosphatase (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Alkaline Phosphatase (U/L)-Day 14 | 61 [50 to 71.5] | 57.5 [53 to 71.5] | 52 [47 to 57] | 48 [42 to 51]
  Alkaline Phosphatase (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Alkaline Phosphatase (U/L)-Day 42 | 55.5 [49 to 73] | 61 [50 to 72] | 51 [45 to 66] | 50 [42 to 64]
  Alkaline Phosphatase (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  Alkaline Phosphatase (U/L)-Day 98 | 54 [49 to 72] | 55 [49 to 70] | 51 [43 to 61] | 52 [44 to 65]
  Alkaline Phosphatase (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  Alkaline Phosphatase (U/L)-Day 182 | 59 [47 to 70] | 56 [48 to 74] | 55 [48 to 67] | 61.5 [56 to 67]
  Alkaline Phosphatase (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Alkaline Phosphatase (U/L)-Day 273 | 57 [50 to 64] | 55 [52.5 to 66] | 53.5 [46 to 61] | 51 [44 to 53]
  creatine phosphokinase (U/L)- Screening | 94 [64 to 130] | 92 [70 to 150] | 88 [61 to 199] | 88 [82 to 269]
  creatine phosphokinase (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  creatine phosphokinase (U/L)-Day 14 | 113.5 [76 to 158] | 92.5 [78 to 123.5] | 58.5 [51 to 66] | 116 [91 to 231]
  creatine phosphokinase (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  creatine phosphokinase (U/L)-Day 42 | 118 [78 to 150] | 91 [69 to 116] | 77 [55 to 135] | 222 [88 to 931]
  creatine phosphokinase (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  creatine phosphokinase (U/L)-Day 98 | 110 [76 to 202] | 102 [68 to 198] | 63 [47 to 75] | 157 [74 to 188]
  creatine phosphokinase (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  creatine phosphokinase (U/L)-Day 182 | 121 [71 to 170] | 99 [69 to 127] | 79 [52 to 89] | 133 [94 to 172]
  creatine phosphokinase (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  creatine phosphokinase (U/L)-Day 273 | 123 [75 to 219] | 98.5 [79 to 175] | 54.5 [47 to 62] | 111 [56 to 224]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in g/dL
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population
Time Frame: Measured during screening, Days 14, 42, 98, 182 and 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
g/dL
  Creatinine (g/dL)- Screening | 0.00084 [0.00077 to 0.00103] | 0.0008 [0.00073 to 0.00087] | 0.00072 [0.00071 to 0.00085] | 0.00093 [0.00073 to 0.00095]
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Creatinine (g/dL)-Day 14 | 0.00086 [0.00074 to 0.001] | 0.00084 [0.00076 to 0.00094] | 0.000645 [0.00061 to 0.00068] | 0.00085 [0.00074 to 0.00095]
  Creatinine (g/dL)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Creatinine (g/dL)-Day 42 | 0.00083 [0.00076 to 0.000975] | 0.00085 [0.00075 to 0.00092] | 0.00072 [0.00059 to 0.00076] | 0.00089 [0.00078 to 0.00094]
  Creatinine (g/dL)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  Creatinine (g/dL)-Day 98 | 0.00085 [0.00076 to 0.00096] | 0.00085 [0.00077 to 0.00091] | 0.00065 [0.00059 to 0.00085] | 0.00093 [0.00077 to 0.001]
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  Creatinine (g/dL)-Day 182 | 0.00084 [0.00077 to 0.00096] | 0.00085 [0.00078 to 0.00092] | 0.00073 [0.00068 to 0.00073] | 0.00081 [0.00074 to 0.00088]
  Creatinine (g/dL)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Creatinine (g/dL)-Day 273 | 0.00088 [0.00081 to 0.00098] | 0.00083 [0.00074 to 0.000895] | 0.00073 [0.00072 to 0.00074] | 0.00084 [0.00081 to 0.00095]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 5
Time Frame: Measured during screening, Days 14, 42, 98, 182 and 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
g/dL
  Hemoglobin (g/dL)- Screening | 14.2 [13.4 to 15] | 14.4 [13.8 to 15.4] | 12.6 [12.1 to 15] | 14.7 [13.5 to 15.4]
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Hemoglobin (g/dL)-Day 14 | 13.8 [12.5 to 15.05] | 13.95 [13.15 to 14.85] | 13.35 [12.3 to 14.4] | 13.9 [12.5 to 14.7]
  Hemoglobin (g/dL)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Hemoglobin (g/dL)-Day 42 | 14.05 [12.7 to 15] | 14 [13 to 14.7] | 12.7 [12.6 to 13.6] | 14.6 [13.1 to 14.9]
  Hemoglobin (g/dL)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Hemoglobin (g/dL)-Day 98 | 14.25 [12.9 to 14.9] | 13.95 [13.2 to 14.7] | 12 [11.9 to 14.1] | 14.6 [11.7 to 15.1]
  Hemoglobin (g/dL)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Hemoglobin (g/dL)-Day 175 | 13.95 [13.3 to 15.1] | 13.45 [12.8 to 14.9] | 13.4 [12.8 to 14.8] | 13.5 [11.8 to 14.9]
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 182 | 12 [11.6 to 12.4] |  |  |
  Hemoglobin (g/dL)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Hemoglobin (g/dL)-Day 273 | 14 [12.7 to 14.7] | 14 [12.65 to 14.6] | 14 [13.2 to 14.8] | 14.6 [11.2 to 15]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count in 1000*Cells/mm^3
Description: as for outcome 5
Time Frame: Measured during screening, Days 14, 42, 98, 175 and 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000*cells/mm^3
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
1000*cells/mm^3
  Neutrophils (1000*cells/mm^3)- Screening | 3.621 [2.507 to 4.458] | 3.564 [2.688 to 4.614] | 3.16 [2.411 to 9.216] | 3.306 [2.981 to 4.061]
  Neutrophils (1000*cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Neutrophils (1000*cells/mm^3)-Day 14 | 3.5165 [2.4525 to 4.196] | 3.1235 [2.347 to 4.678] | 5.1805 [3.959 to 6.402] | 3.224 [2.91 to 4.044]
  Neutrophils (1000*cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Neutrophils (1000*cells/mm^3)-Day 42 | 3.348 [2.4 to 4.1765] | 3.036 [2.671 to 3.917] | 2.292 [1.436 to 5.035] | 3.31 [3.042 to 4.522]
  Neutrophils (1000*cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Neutrophils (1000*cells/mm^3)-Day 98 | 2.9925 [2.723 to 3.522] | 3.0915 [2.539 to 3.892] | 2.961 [2.744 to 5.623] | 2.626 [2.158 to 3.859]
  Neutrophils (1000*cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Neutrophils (1000*cells/mm^3)-Day 175 | 2.773 [2.244 to 3.119] | 2.7645 [2.22 to 3.673] | 2.902 [1.742 to 3.688] | 4.694 [2.979 to 6.17]
  Neutrophils (1000*cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Neutrophils (1000*cells/mm^3)-Day 182 | 3.018 [2.298 to 3.738] |  |  |
  Neutrophils (1000*cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Neutrophils (1000*cells/mm^3)-Day 273 | 3.279 [2.654 to 3.81] | 3.011 [2.346 to 3.859] | 6.428 [1.76 to 11.096] | 2.677 [1.901 to 2.783]
  Lymphocytes (1000*cells/mm^3)- Screening | 1.916 [1.47 to 2.09] | 1.765 [1.4 to 2.18] | 1.84 [1.2 to 2.757] | 1.928 [1.904 to 2.74]
  Lymphocytes (1000*cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Lymphocytes (1000*cells/mm^3)-Day 14 | 1.907 [1.5705 to 2.269] | 1.873 [1.6115 to 2.3815] | 2.9485 [2.3 to 3.597] | 1.712 [1.5 to 1.83]
  Lymphocytes (1000*cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Lymphocytes (1000*cells/mm^3)-Day 42 | 1.8925 [1.5395 to 2.245] | 1.88 [1.51 to 2.26] | 2.35 [0.86 to 3.216] | 2.037 [1.986 to 2.09]
  Lymphocytes (1000*cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Lymphocytes (1000*cells/mm^3)-Day 98 | 1.8265 [1.503 to 2.211] | 1.668 [1.464 to 2.244] | 2.13 [1.07 to 2.744] | 2.15 [1.786 to 3.441]
  Lymphocytes (1000*cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Lymphocytes (1000*cells/mm^3)-Day 175 | 1.8365 [1.66 to 2.251] | 1.846 [1.472 to 2.14] | 1.42 [0.91 to 2.917] | 1.855 [1.793 to 3.25]
  Lymphocytes (1000*cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Lymphocytes (1000*cells/mm^3)-Day 182 | 1.847 [1.824 to 1.87] |  |  |
  Lymphocytes (1000*cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Lymphocytes (1000*cells/mm^3)-Day 273 | 1.717 [1.587 to 2.009] | 1.701 [1.45 to 2.0205] | 1.76 [0.89 to 2.63] | 2.328 [1.651 to 2.37]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC in 1000*Cells/mm^3
Description: as for outcome 5
Time Frame: Measured during screening, Days 14, 42, 98, 175 and 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000*cells/mm^3
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
1000*cells/mm^3
  WBC (1000*cells/mm^3)- Screening | 6.2 [5 to 6.7] | 6.4 [5.2 to 7.5] | 7.9 [4.2 to 12] | 5.7 [5.4 to 7.2]
  WBC (1000*cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  WBC (1000*cells/mm^3)-Day 14 | 6.25 [5.3 to 7.05] | 5.55 [4.85 to 7.45] | 9.75 [9.7 to 9.8] | 5.4 [5.3 to 6]
  WBC (1000*cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  WBC (1000*cells/mm^3)-Day 42 | 6 [4.85 to 7.05] | 6 [4.8 to 6.8] | 8.1 [2.8 to 8.2] | 5.9 [5.5 to 7]
  WBC (1000*cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  WBC (1000*cells/mm^3)-Day 98 | 5.75 [5 to 6.3] | 5.35 [4.5 to 6.9] | 7 [4.5 to 8.8] | 6.2 [4.8 to 6.4]
  WBC (1000*cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  WBC (1000*cells/mm^3)-Day 175 | 5.3 [4.9 to 5.9] | 5.1 [4.5 to 6.8] | 5.9 [3.1 to 7.8] | 7.2 [5.3 to 10]
  WBC (1000*cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  WBC (1000*cells/mm^3)-Day 182 | 5.45 [4.9 to 6] |  |  |
  WBC (1000*cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  WBC (1000*cells/mm^3)-Day 273 | 5.9 [5.1 to 6.5] | 5.55 [4.4 to 6.75] | 8.9 [3.2 to 14.6] | 4.9 [4.8 to 5.6]
  Platelets (1000*cells/mm^3)- Screening | 271 [236 to 305] | 244 [198 to 294] | 274 [206 to 347] | 264 [213 to 276]
  Platelets (1000*cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Platelets (1000*cells/mm^3)-Day 14 | 276.5 [241.5 to 301] | 269 [241 to 330] | 335 [292 to 378] | 231 [213 to 254]
  Platelets (1000*cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Platelets (1000*cells/mm^3)-Day 42 | 261.5 [242.5 to 297.5] | 260 [238 to 300] | 265 [225 to 402] | 226 [226 to 239]
  Platelets (1000*cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Platelets (1000*cells/mm^3)-Day 98 | 275 [255 to 292] | 241 [207 to 306] | 302 [203 to 394] | 262 [226 to 266]
  Platelets (1000*cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Platelets (1000*cells/mm^3)-Day 175 | 271 [242 to 292] | 241.5 [215 to 260] | 255 [243 to 352] | 256 [224 to 269]
  Platelets (1000*cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Platelets (1000*cells/mm^3)-Day 182 | 255.5 [246 to 265] |  |  |
  Platelets (1000*cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Platelets (1000*cells/mm^3)-Day 273 | 284 [233 to 306] | 243.5 [217 to 279] | 229.5 [223 to 236] | 232 [219 to 263]

9. Primary Outcome: Number of Participants With Chemistry and Hematology Laboratory Measures - Counts of Lab Grade > 1
Description: The number (percentage) of participants with Chemistry and Hematology Laboratory Measures - Counts of Lab Grade > 1 for alkaline phosphate (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatine phosphokinase (CPK), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by treatment group and visit time
Time Frame: Measured during screening, Days 14, 42, 98, 182 and 273 for (ALP), (AST), (ALT), (CPK), creatinine. Measured during screening, Days 14, 42, 98, 175, 182 and 273 for Lymphocyte count, Neutrophil count Platelets, WBC, hemoglobin.
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit. Visit schedule is not the same for each laboratory measures. For visits not on the schedule, number analyzed is 0 or applicable participants number.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  WBC (1000*Cells/mm^3)- Screening | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  WBC (1000*Cells/mm^3)-Day 14 | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  WBC (1000*Cells/mm^3)-Day 42 | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  WBC (1000*Cells/mm^3)-Day 98 | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  WBC (1000*Cells/mm^3)-Day 175 | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 182 | 0 | 0 | 0 | 0
  WBC (1000*Cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  WBC (1000*Cells/mm^3)-Day 273 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)- Screening | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Neutrophils (1000*Cells/mm^3)-Day 14 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Neutrophils (1000*Cells/mm^3)-Day 42 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Neutrophils (1000*Cells/mm^3)-Day 98 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Neutrophils (1000*Cells/mm^3)-Day 175 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 182 | 0 | 0 | 0 | 0
  Neutrophils (1000*Cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Neutrophils (1000*Cells/mm^3)-Day 273 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Screening | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Hemoglobin (g/dL)-Day 14 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Hemoglobin (g/dL)-Day 42 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Hemoglobin (g/dL)-Day 98 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Hemoglobin (g/dL)-Day 175 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 182 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Hemoglobin (g/dL)-Day 273 | 1 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)- Screening | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Lymphocytes (1000*Cells/mm^3)-Day 14 | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Lymphocytes (1000*Cells/mm^3)-Day 42 | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Lymphocytes (1000*Cells/mm^3)-Day 98 | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Lymphocytes (1000*Cells/mm^3)-Day 175 | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 182 | 0 | 0 | 0 | 0
  Lymphocytes (1000*Cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Lymphocytes (1000*Cells/mm^3)-Day 273 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)- Screening | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Platelets (1000*Cells/mm^3)-Day 14 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Platelets (1000*Cells/mm^3)-Day 42 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 98: number analyzed (Participants) | 22 | 22 | 3 | 3
  Platelets (1000*Cells/mm^3)-Day 98 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 175: number analyzed (Participants) | 18 | 22 | 3 | 3
  Platelets (1000*Cells/mm^3)-Day 175 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 182: number analyzed (Participants) | 2 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 182 | 0 | 0 | 0 | 0
  Platelets (1000*Cells/mm^3)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Platelets (1000*Cells/mm^3)-Day 273 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Screening | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  ALT (SGPT) (U/L)-Day 14 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  ALT (SGPT) (U/L)-Day 42 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  ALT (SGPT) (U/L)-Day 98 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 175 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  ALT (SGPT) (U/L)-Day 182 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  ALT (SGPT) (U/L)-Day 273 | 0 | 0 | 0 | 0
  AST (U/L)- Screening | 0 | 0 | 0 | 0
  AST (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  AST (U/L)-Day 14 | 0 | 0 | 0 | 0
  AST (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  AST (U/L)-Day 42 | 0 | 0 | 0 | 0
  AST (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  AST (U/L)-Day 98 | 0 | 0 | 0 | 0
  AST (U/L)-Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST (U/L)-Day 175 | 0 | 0 | 0 | 0
  AST (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  AST (U/L)-Day 182 | 0 | 0 | 0 | 0
  AST (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 2
  AST (U/L)-Day 273 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Screening | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Alkaline Phosphatase (U/L)-Day 14 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Alkaline Phosphatase (U/L)-Day 42 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  Alkaline Phosphatase (U/L)-Day 98 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 175 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  Alkaline Phosphatase (U/L)-Day 182 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Alkaline Phosphatase (U/L)-Day 273 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Screening | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  Creatinine (g/dL)-Day 14 | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  Creatinine (g/dL)-Day 42 | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  Creatinine (g/dL)-Day 98 | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 175 | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  Creatinine (g/dL)-Day 182 | 0 | 0 | 0 | 0
  Creatinine (g/dL)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  Creatinine (g/dL)-Day 273 | 0 | 1 | 0 | 0
  creatine phosphokinase (U/L)- Screening | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 14: number analyzed (Participants) | 24 | 24 | 2 | 3
  creatine phosphokinase (U/L)-Day 14 | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 42: number analyzed (Participants) | 24 | 25 | 3 | 3
  creatine phosphokinase (U/L)-Day 42 | 0 | 0 | 0 | 1
  creatine phosphokinase (U/L)-Day 98: number analyzed (Participants) | 22 | 23 | 3 | 3
  creatine phosphokinase (U/L)-Day 98 | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 175 | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 182: number analyzed (Participants) | 23 | 23 | 3 | 2
  creatine phosphokinase (U/L)-Day 182 | 0 | 0 | 0 | 0
  creatine phosphokinase (U/L)-Day 273: number analyzed (Participants) | 21 | 24 | 2 | 3
  creatine phosphokinase (U/L)-Day 273 | 0 | 2 | 0 | 0

10. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  Refused study product administration | 3 | 1 | 0 | 1
  Clinical event (not reacto, HIV, death) | 1 | 1 | 0 | 0
  Investigator decision | 1 | 0 | 0 | 0
  EP device difficulty | 0 | 1 | 0 | 0
  Participant Relocated | 0 | 1 | 0 | 0
  Did not discontinue SPA | 20 | 21 | 3 | 2

11. Primary Outcome: Magnitude of Local Injection/EP Site Pain as Measured by a Visual Analog Scale (Day 0, Day 28, Day 84, Day 168)
Description: A visual analog scale is a horizontal line, 10 cm in length, anchored by word descriptors at each end ("no pain" and "worst pain"). The visual analog scale score is determined by measuring in centimeters from the left hand end of the line to the point that the patient marks, 0 cm being no pain and 10 cm being maximum pain.The pain assessment scores for each arm at each vaccination visit were summarized with visual analog scale (VAS)
Time Frame: Measured during Day 0, 28, 84 and 168
Population: One participant in Group 1 had VASOVAGAL REACTION AND SEIZURE on enrollment visit. One participant in Group 2 experienced EP device difficulty on enrollment visit. These two participants had no Visual Analog Scale - Pain Assessment Scores.
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Score
  0 - V2.0 - Day 0: number analyzed (Participants) | 24 | 24 | 3 | 3
  0 - V2.0 - Day 0 | 4.65 [2.1 to 7.05] | 4.75 [1.9 to 6.4] | 6.9 [4.4 to 7.9] | 4.9 [0.6 to 8.4]
  5-7 - V2.0 - Day 0: number analyzed (Participants) | 24 | 24 | 3 | 3
  5-7 - V2.0 - Day 0 | 0.8 [0 to 1.95] | 0.85 [0.2 to 2.05] | 2.2 [0.5 to 4.7] | 1.7 [0.3 to 1.8]
  25_60 - V2.0 - Day 0: number analyzed (Participants) | 24 | 24 | 3 | 3
  25_60 - V2.0 - Day 0 | 0.45 [0 to 1.4] | 0.7 [0.1 to 1.1] | 1.7 [0.3 to 2.1] | 0.7 [0.3 to 1.8]
  0 - V4.0 - Day 28: number analyzed (Participants) | 22 | 22 | 3 | 2
  0 - V4.0 - Day 28 | 4.3 [3.2 to 6.9] | 3.65 [1.4 to 5.5] | 5.5 [3.7 to 6.4] | 3.3 [3.1 to 3.5]
  5-7 - V4.0 - Day 28: number analyzed (Participants) | 22 | 23 | 3 | 2
  5-7 - V4.0 - Day 28 | 1.6 [0.9 to 2.8] | 0.7 [0.2 to 2.2] | 2.4 [1.8 to 4.2] | 1.05 [1 to 1.1]
  25_60 - V4.0 - Day 28: number analyzed (Participants) | 22 | 23 | 3 | 2
  25_60 - V4.0 - Day 28 | 0.5 [0.3 to 1.2] | 0.5 [0.2 to 1.4] | 1.8 [1 to 3.6] | 0.65 [0.3 to 1]
  0 - V7.0 - Day 84: number analyzed (Participants) | 22 | 21 | 2 | 2
  0 - V7.0 - Day 84 | 3.95 [3.1 to 6.9] | 3.6 [1.8 to 4.9] | 6.85 [4.4 to 9.3] | 5 [2.2 to 7.8]
  5-7 - V7.0 - Day 84: number analyzed (Participants) | 22 | 21 | 2 | 2
  5-7 - V7.0 - Day 84 | 1.1 [0.2 to 1.8] | 0.8 [0.2 to 1.2] | 1.7 [1.6 to 1.8] | 2.15 [0.4 to 3.9]
  25_60 - V7.0 - Day 84: number analyzed (Participants) | 22 | 21 | 2 | 2
  25_60 - V7.0 - Day 84 | 0.55 [0.1 to 0.9] | 0.3 [0 to 0.9] | 1.1 [1 to 1.2] | 1.9 [0.2 to 3.6]
  0 - V9.0 - Day 168: number analyzed (Participants) | 19 | 20 | 1 | 2
  0 - V9.0 - Day 168 | 5.1 [1.5 to 6.8] | 3.95 [0.4 to 5.75] | 3.4 [3.4 to 3.4] | 2.6 [0.7 to 4.5]
  5-7 - V9.0 - Day 168: number analyzed (Participants) | 19 | 20 | 1 | 2
  5-7 - V9.0 - Day 168 | 0.8 [0.1 to 1.6] | 0.6 [0.1 to 2] | 2.4 [2.4 to 2.4] | 0.75 [0.5 to 1]
  25_60 - V9.0 - Day 168: number analyzed (Participants) | 19 | 20 | 1 | 2
  25_60 - V9.0 - Day 168 | 0.2 [0.1 to 0.5] | 0.3 [0 to 1] | 0.8 [0.8 to 0.8] | 0.3 [0.2 to 0.4]

12. Primary Outcome: Distribution of Responses to Questions Regarding Acceptability of Study Injection Procedures [ Visits 3, 5, 8, 10]
Description: Distribution of responses to questions regarding acceptability of study injection procedures [ Visits 3, 5, 8, 10] were summarized by category (Acceptable/Unacceptable/Don?t know/ Don?t Remember)
Time Frame: Measured during Visit 3 (Day14), Visit 5 (Day 35), Visit 8 (Day 98), Visit 10 (Day 175)
Population: One participant in Group 1 had VASOVAGAL REACTION AND SEIZURE on enrollment. One participant in Group 2 had an interim visit done as the visit was done prior to the visit 3.0 window opening. Data Manager instructed site to complete the interim visit and then following w/ a missed visit. These two cases were missed in the enrollment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 3 | 3
Participants
  Question-1- Acceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-1- Acceptable- Day 14 | 17 | 20 | 3 | 2
  Question-1- Unacceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-1- Unacceptable- Day 14 | 7 | 2 | 0 | 1
  Question-1- Don't Know/Don't Remember- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-1- Don't Know/Don't Remember- Day 14 | 0 | 2 | 0 | 0
  Question-1- Acceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-1- Acceptable- Day 175 | 16 | 19 | 3 | 2
  Question-1- Unacceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-1- Unacceptable- Day 175 | 2 | 2 | 0 | 0
  Question-1- Don't Know/Don't Remember- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-1- Don't Know/Don't Remember- Day 175 | 0 | 0 | 0 | 0
  Question-1- Acceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-1- Acceptable- Day 35 | 20 | 20 | 3 | 2
  Question-1- Unacceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-1- Unacceptable- Day 35 | 3 | 2 | 0 | 0
  Question-1- Don't Know/Don't Remember- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-1- Don't Know/Don't Remember- Day 35 | 0 | 0 | 0 | 0
  Question-1- Acceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-1- Acceptable- Day 98 | 19 | 18 | 3 | 2
  Question-1- Unacceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-1- Unacceptable- Day 98 | 3 | 3 | 0 | 0
  Question-1- Don't Know/Don't Remember- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-1- Don't Know/Don't Remember- Day 98 | 0 | 1 | 0 | 0
  Question-2- Acceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-2- Acceptable- Day 14 | 22 | 23 | 3 | 3
  Question-2- Unacceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-2- Unacceptable- Day 14 | 2 | 0 | 0 | 0
  Question-2- Don't Know/Don't Remember- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-2- Don't Know/Don't Remember- Day 14 | 0 | 1 | 0 | 0
  Question-2- Acceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-2- Acceptable- Day 175 | 17 | 21 | 3 | 2
  Question-2- Unacceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-2- Unacceptable- Day 175 | 1 | 0 | 0 | 0
  Question-2- Don't Know/Don't Remember- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-2- Don't Know/Don't Remember- Day 175 | 0 | 0 | 0 | 0
  Question-2- Acceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-2- Acceptable- Day 35 | 22 | 20 | 3 | 2
  Question-2- Unacceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-2- Unacceptable- Day 35 | 1 | 2 | 0 | 0
  Question-2- Don't Know/Don't Remember- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-2- Don't Know/Don't Remember- Day 35 | 0 | 0 | 0 | 0
  Question-2- Acceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-2- Acceptable- Day 98 | 20 | 21 | 3 | 2
  Question-2- Unacceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-2- Unacceptable- Day 98 | 2 | 0 | 0 | 0
  Question-2- Don't Know/Don't Remember- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-2- Don't Know/Don't Remember- Day 98 | 0 | 1 | 0 | 0
  Question-3- Acceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-3- Acceptable- Day 14 | 19 | 21 | 2 | 3
  Question-3- Unacceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-3- Unacceptable- Day 14 | 4 | 2 | 1 | 0
  Question-3- Don't Know/Don't Remember- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-3- Don't Know/Don't Remember- Day 14 | 1 | 1 | 0 | 0
  Question-3- Acceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-3- Acceptable- Day 175 | 15 | 18 | 1 | 2
  Question-3- Unacceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-3- Unacceptable- Day 175 | 3 | 3 | 0 | 0
  Question-3- Don't Know/Don't Remember- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-3- Don't Know/Don't Remember- Day 175 | 0 | 0 | 2 | 0
  Question-3- Acceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-3- Acceptable- Day 35 | 18 | 19 | 3 | 2
  Question-3- Unacceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-3- Unacceptable- Day 35 | 5 | 3 | 0 | 0
  Question-3- Don't Know/Don't Remember- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-3- Don't Know/Don't Remember- Day 35 | 0 | 0 | 0 | 0
  Question-3- Acceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-3- Acceptable- Day 98 | 20 | 19 | 2 | 2
  Question-3- Unacceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-3- Unacceptable- Day 98 | 2 | 3 | 1 | 0
  Question-3- Don't Know/Don't Remember- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-3- Don't Know/Don't Remember- Day 98 | 0 | 0 | 0 | 0
  Question-4- Acceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-4- Acceptable- Day 14 | 24 | 24 | 3 | 3
  Question-4- Unacceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-4- Unacceptable- Day 14 | 0 | 0 | 0 | 0
  Question-4- Don't Know/Don't Remember- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-4- Don't Know/Don't Remember- Day 14 | 0 | 0 | 0 | 0
  Question-4- Acceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-4- Acceptable- Day 175 | 18 | 20 | 3 | 2
  Question-4- Unacceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-4- Unacceptable- Day 175 | 0 | 1 | 0 | 0
  Question-4- Don't Know/Don't Remember- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-4- Don't Know/Don't Remember- Day 175 | 0 | 0 | 0 | 0
  Question-4- Acceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-4- Acceptable- Day 35 | 23 | 20 | 2 | 2
  Question-4- Unacceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-4- Unacceptable- Day 35 | 0 | 2 | 1 | 0
  Question-4- Don't Know/Don't Remember- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-4- Don't Know/Don't Remember- Day 35 | 0 | 0 | 0 | 0
  Question-4- Acceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-4- Acceptable- Day 98 | 22 | 21 | 3 | 2
  Question-4- Unacceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-4- Unacceptable- Day 98 | 0 | 0 | 0 | 0
  Question-4- Don't Know/Don't Remember- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-4- Don't Know/Don't Remember- Day 98 | 0 | 1 | 0 | 0
  Question-5- Acceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-5- Acceptable- Day 14 | 4 | 8 | 0 | 0
  Question-5- Unacceptable- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-5- Unacceptable- Day 14 | 0 | 0 | 0 | 0
  Question-5- Don't Know/Don't Remember- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-5- Don't Know/Don't Remember- Day 14 | 0 | 1 | 1 | 0
  Question-5- No Other Side Effects- Day 14: number analyzed (Participants) | 24 | 24 | 3 | 3
  Question-5- No Other Side Effects- Day 14 | 20 | 15 | 2 | 3
  Question-5- Acceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-5- Acceptable- Day 175 | 2 | 1 | 0 | 1
  Question-5- Unacceptable- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-5- Unacceptable- Day 175 | 1 | 0 | 0 | 0
  Question-5- Don't Know/Don't Remember- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-5- Don't Know/Don't Remember- Day 175 | 0 | 0 | 0 | 0
  Question-5- No Other Side Effects- Day 175: number analyzed (Participants) | 18 | 21 | 3 | 2
  Question-5- No Other Side Effects- Day 175 | 15 | 20 | 3 | 1
  Question-5- Acceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-5- Acceptable- Day 35 | 4 | 5 | 1 | 0
  Question-5- Unacceptable- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-5- Unacceptable- Day 35 | 0 | 2 | 0 | 0
  Question-5- Don't Know/Don't Remember- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-5- Don't Know/Don't Remember- Day 35 | 0 | 0 | 0 | 0
  Question-5- No Other Side Effects- Day 35: number analyzed (Participants) | 23 | 22 | 3 | 2
  Question-5- No Other Side Effects- Day 35 | 19 | 15 | 2 | 2
  Question-5- Acceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-5- Acceptable- Day 98 | 1 | 4 | 0 | 0
  Question-5- Unacceptable- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-5- Unacceptable- Day 98 | 0 | 1 | 0 | 0
  Question-5- Don't Know/Don't Remember- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-5- Don't Know/Don't Remember- Day 98 | 1 | 1 | 0 | 0
  Question-5- No Other Side Effects- Day 98: number analyzed (Participants) | 22 | 22 | 3 | 2
  Question-5- No Other Side Effects- Day 98 | 20 | 16 | 3 | 2

13. Primary Outcome: Summary of T-Cell Epitope Mapping Breadth (Defined as the Number of Targeted CEs) Among All Participants by T-cell Subset (CD4+, CD8+), Visit, and Treatment Arm [Time Frame: Measured at M1.5 and M6.5]
Description: For participants with a positive Fisher's Exact response to Gag CE Total and/or HBX2 p55Gag for either IFN-γ and/or IL2(CD4+ or CD8+) or for CD40L(CD4+)at month1.5and/or month 6.5, samples were further assayed against the seven individual CE peptide pools and the total number of positive responses was defined as the breadth.
Time Frame: M1.5 and M6.5
Population: Immunogenicity Population. Group 3 and Group 4 are control groups. Control groups were excluded in this analysis because that no peptide responses were expected in control groups. This is pre-specified in Study Analysis Plan.
Measure: Mean (95% Confidence Interval); unit: Number of targeted CEs
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 24 | 25
Number of targeted CEs
  IFNg+ - CD4+ - M1.5: number analyzed (Participants) | 23 | 24
  IFNg+ - CD4+ - M1.5 | 0.261 [0.096 to 0.591] | 0.333 [0.141 to 0.699]
  IFNg+ - CD4+ - M6.5: number analyzed (Participants) | 22 | 23
  IFNg+ - CD4+ - M6.5 | 0.682 [0.375 to 1.159] | 0.217 [0.075 to 0.487]
  IFNg+ - CD8+ - M1.5: number analyzed (Participants) | 24 | 24
  IFNg+ - CD8+ - M1.5 | 0.042 [NA to NA] — Negative binomial regression failed to estimated the variance due to over-dispersion parameter when applied. | 0.25 [NA to NA] — Negative binomial regression failed to estimated the variance due to over-dispersion parameter when applied.
  IFNg+ - CD8+ - M6.5: number analyzed (Participants) | 22 | 23
  IFNg+ - CD8+ - M6.5 | 0.455 [0.215 to 0.87] | 0.304 [0.125 to 0.634]
  IFNg+ - Overall - M1.5: number analyzed (Participants) | 23 | 24
  IFNg+ - Overall - M1.5 | 0.304 [0.12 to 0.672] | 0.583 [0.295 to 1.109]
  IFNg+ - Overall - M6.5: number analyzed (Participants) | 22 | 23
  IFNg+ - Overall - M6.5 | 1.136 [0.697 to 1.801] | 0.522 [0.267 to 0.936]

14. Secondary Outcome: CD4+ and CD8+ T Cell Response Rate Measured by Flow Cytometry to p24CE and HIV Gag by Cytokine, T-cell Subset (CD4+, CD8+), Antigen and Treatment Group [Time Frame: Measured at M0, M1.5 and M6.5]
Description: Flow cytometry was used to examine HIV-1 specific CD4+ and CD8+ T-cell responses using a validated ICS assay. A one sided Fisher's exact test was applied to detective the positivity response. If at least one peptide pool for a specific HIV-1 protein was positive, then the overall response to the protein was considered positive. If any peptide pool was positive for a T-cellubset, then the overall response for that T-cell subset was considered positive.
Time Frame: M0, M1.5 and M6.5
Population: Immunogenicity Population
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: Control 1 + Group 4: Control 2: Placebo: Sodium Chloride, USP 0.9%
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 + Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 6
Participants
  CD40L+ - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5 | 8 | 7 | 0
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5 | 15 | 9 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5 | 9 | 22 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5 | 20 | 21 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5 | 7 | 8 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5 | 14 | 8 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5 | 7 | 22 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5 | 20 | 19 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 24 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5 | 1 | 5 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5 | 9 | 5 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 24 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5 | 1 | 9 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5 | 5 | 16 | 0

15. Secondary Outcome: CD4+ and CD8+ T Cell MIMOSA Response Rate Measured by Flow Cytometry to p24CE and HIV Gag by Cytokine, T-cell Subset (CD4+, CD8+), Antigen and Treatment Group [Time Frame: Measured at M0, M1.5 and M6.5]
Description: Flow cytometry was used to examine HIV-1 specific CD4+ and CD8+ T-cell responses using a validated ICS assay. Athe Mixture Models for Single-cell Assays (MIMOSA) statistical framework was applied to detective the positivity response. If at least one peptide pool for a specific HIV-1 protein was positive, then the overall response to the protein was considered positive. If any peptide pool was positive for a T-cellubset, then the overall response for that T-cell subset was considered positive.
Time Frame: M0, M1.5 and M6.5
Population: Immunogenicity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 + Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 6
Participants
  CD40L+ - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5 | 8 | 8 | 0
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5 | 16 | 11 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5 | 9 | 22 | 0
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5 | 20 | 22 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5 | 7 | 8 | 0
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5 | 14 | 9 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5 | 8 | 22 | 0
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5 | 20 | 19 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 24 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5 | 1 | 5 | 0
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5 | 9 | 5 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 24 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0 | 0 | 0 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5 | 1 | 10 | 0
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5 | 5 | 18 | 0

16. Secondary Outcome: Summary of CD4+ and CD8+ T Cell Response Magnitudes Among All Participants by Cytokine, T-Cell Subset (CD4+, CD8+), Antigen and Treatment Group [Time Frame: Measured at M0, M1.5 and M6.5]
Description: Flow cytometry was used to examine HIV-1 specific CD4+ and CD8+ T-cell responses using a validated ICS assay. Percentage of CD4+ T cells expressing CD40L+ was used as the magnititudes response for ICS assay.
Time Frame: M0, M1.5 and M6.5
Population: Immunogenicity Population
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 + Group 4: Control 2
Number analyzed (Participants) | 25 | 25 | 6
percentage
  CD40L+ - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 1.5 | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0]
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - Gag CE Total - at Month 6.5 | 0.1 [0.1 to 0.2] | 0 [0 to 0.1] | 0 [0 to 0]
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 24 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 1.5 | 0 [0 to 0.1] | 0.3 [0.2 to 0.3] | 0 [0 to 0]
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  CD40L+ - CD4+ - HBX2 p55 Gag - at Month 6.5 | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 25 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 1.5 | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - Gag CE Total - at Month 6.5 | 0.1 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 25 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 24 | 23 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 1.5 | 0 [0 to 0.1] | 0.3 [0.2 to 0.4] | 0 [0 to 0]
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 21 | 6
  IFNg/IL2 - CD4+ - HBX2 p55 Gag - at Month 6.5 | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.4] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0: number analyzed (Participants) | 20 | 24 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 1.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - Gag CE Total - at Month 6.5 | 0 [0 to 0.2] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0: number analyzed (Participants) | 22 | 24 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5: number analyzed (Participants) | 23 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 1.5 | 0 [0 to 0] | 0.1 [0 to 0.2] | 0 [0 to 0]
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5: number analyzed (Participants) | 22 | 23 | 6
  IFNg/IL2 - CD8+ - HBX2 p55 Gag - at Month 6.5 | 0 [0 to 0] | 0.1 [0.1 to 0.5] | 0 [0 to 0]

17. Secondary Outcome: CD4+ and CD8+ T Cell Response Rate Measured by Flow Cytometry to p24CE and HIV Gag by Cytokine, T-cell Subset (CD4+, CD8+), Antigen and Treatment Group [Time Frame: Measured at M1.5 and M6.5]
Description: as for outcome 14
Time Frame: M0, M1.5 and M6.5
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 24 | 25
Participants
  IFNg+ - CD4+ - Gag CE 1 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 1 - M1.5 | 0 | 4
  IFNg+ - CD4+ - Gag CE 1 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 1 - M6.5 | 1 | 2
  IFNg+ - CD4+ - Gag CE 2 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 2 - M1.5 | 0 | 0
  IFNg+ - CD4+ - Gag CE 2 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD4+ - Gag CE 2 - M6.5 | 1 | 0
  IFNg+ - CD4+ - Gag CE 3 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 3 - M1.5 | 1 | 0
  IFNg+ - CD4+ - Gag CE 3 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 3 - M6.5 | 1 | 0
  IFNg+ - CD4+ - Gag CE 4 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 4 - M1.5 | 0 | 0
  IFNg+ - CD4+ - Gag CE 4 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 4 - M6.5 | 0 | 0
  IFNg+ - CD4+ - Gag CE 5 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 5 - M1.5 | 3 | 1
  IFNg+ - CD4+ - Gag CE 5 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 5 - M6.5 | 6 | 0
  IFNg+ - CD4+ - Gag CE 6 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 6 - M1.5 | 2 | 3
  IFNg+ - CD4+ - Gag CE 6 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 6 - M6.5 | 6 | 3
  IFNg+ - CD4+ - Gag CE 7 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 7 - M1.5 | 0 | 0
  IFNg+ - CD4+ - Gag CE 7 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD4+ - Gag CE 7 - M6.5 | 0 | 0
  IFNg+ - CD4+ - Gag p15 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag p15 - M1.5 | 0 | 9
  IFNg+ - CD4+ - Gag p15 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p15 - M6.5 | 3 | 9
  IFNg+ - CD4+ - Gag p17 - M1.5: number analyzed (Participants) | 9 | 21
  IFNg+ - CD4+ - Gag p17 - M1.5 | 0 | 18
  IFNg+ - CD4+ - Gag p17 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p17 - M6.5 | 6 | 14
  IFNg+ - CD4+ - Gag p24 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag p24 - M1.5 | 6 | 18
  IFNg+ - CD4+ - Gag p24 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p24 - M6.5 | 17 | 14
  IFNg+ - CD8+ - Gag CE 1 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 1 - M1.5 | 0 | 0
  IFNg+ - CD8+ - Gag CE 1 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 1 - M6.5 | 2 | 0
  IFNg+ - CD8+ - Gag CE 2 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 2 - M1.5 | 0 | 1
  IFNg+ - CD8+ - Gag CE 2 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD8+ - Gag CE 2 - M6.5 | 1 | 0
  IFNg+ - CD8+ - Gag CE 3 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 3 - M1.5 | 0 | 3
  IFNg+ - CD8+ - Gag CE 3 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 3 - M6.5 | 1 | 2
  IFNg+ - CD8+ - Gag CE 4 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 4 - M1.5 | 1 | 2
  IFNg+ - CD8+ - Gag CE 4 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 4 - M6.5 | 3 | 3
  IFNg+ - CD8+ - Gag CE 5 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 5 - M1.5 | 0 | 1
  IFNg+ - CD8+ - Gag CE 5 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 5 - M6.5 | 1 | 1
  IFNg+ - CD8+ - Gag CE 6 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 6 - M1.5 | 0 | 1
  IFNg+ - CD8+ - Gag CE 6 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 6 - M6.5 | 2 | 1
  IFNg+ - CD8+ - Gag CE 7 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 7 - M1.5 | 0 | 0
  IFNg+ - CD8+ - Gag CE 7 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD8+ - Gag CE 7 - M6.5 | 0 | 0
  IFNg+ - CD8+ - Gag p15 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag p15 - M1.5 | 0 | 3
  IFNg+ - CD8+ - Gag p15 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p15 - M6.5 | 0 | 3
  IFNg+ - CD8+ - Gag p17 - M1.5: number analyzed (Participants) | 9 | 21
  IFNg+ - CD8+ - Gag p17 - M1.5 | 0 | 2
  IFNg+ - CD8+ - Gag p17 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p17 - M6.5 | 0 | 3
  IFNg+ - CD8+ - Gag p24 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag p24 - M1.5 | 1 | 4
  IFNg+ - CD8+ - Gag p24 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p24 - M6.5 | 7 | 7

18. Secondary Outcome: Summary of CD4+ and CD8+ T Cell Response Magnitudes to Epitope Mapping Gag Among All Participants by by Cytokine, T-Cell Subset (CD4+, CD8+), Antigenand Treatment Group [Time Frame: Measured at M1.5 and M6.5]
Description: For participants with a positive Fisher's Exact response to Gag CE Total and/or HBX2 p55Gag for either IFN-γ and/or IL2(CD4+ or CD8+) or for CD40L(CD4+)at month1.5and/or month 6.5, samples were further assayed against the seven individual CE peptide pools. Percentage of CD8+ T cells expressing IFN-gamma was used as the magnitude response. The background-substracted magnitude was summarized by treatment group. The negative reading of magnitude is due to background substracted.
Time Frame: M1.5 and M6.5
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 22 | 24
percentage
  IFNg+ - CD4+ - Gag CE 1 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 1 - M1.5 | -0.003 [-0.004 to -0.001] | 0.002 [-0.002 to 0.007]
  IFNg+ - CD4+ - Gag CE 1 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 1 - M6.5 | -0.002 [-0.005 to 0.002] | 0.003 [-0.003 to 0.007]
  IFNg+ - CD4+ - Gag CE 2 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 2 - M1.5 | 0 [-0.003 to 0.002] | 0.001 [-0.003 to 0.004]
  IFNg+ - CD4+ - Gag CE 2 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD4+ - Gag CE 2 - M6.5 | -0.001 [-0.004 to 0.01] | 0.002 [-0.003 to 0.005]
  IFNg+ - CD4+ - Gag CE 3 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 3 - M1.5 | 0 [-0.003 to 0.007] | 0 [-0.002 to 0.003]
  IFNg+ - CD4+ - Gag CE 3 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 3 - M6.5 | -0.001 [-0.004 to 0.007] | -0.001 [-0.004 to 0.004]
  IFNg+ - CD4+ - Gag CE 4 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 4 - M1.5 | 0.001 [0 to 0.007] | 0.002 [-0.001 to 0.005]
  IFNg+ - CD4+ - Gag CE 4 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 4 - M6.5 | 0.002 [-0.004 to 0.005] | 0.001 [-0.002 to 0.007]
  IFNg+ - CD4+ - Gag CE 5 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 5 - M1.5 | 0.034 [0.017 to 0.043] | 0.005 [0.002 to 0.01]
  IFNg+ - CD4+ - Gag CE 5 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 5 - M6.5 | 0.022 [0.015 to 0.035] | 0.002 [-0.002 to 0.008]
  IFNg+ - CD4+ - Gag CE 6 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 6 - M1.5 | 0.008 [0 to 0.024] | 0.012 [0.002 to 0.02]
  IFNg+ - CD4+ - Gag CE 6 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag CE 6 - M6.5 | 0.02 [0.005 to 0.039] | 0.004 [0.001 to 0.016]
  IFNg+ - CD4+ - Gag CE 7 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag CE 7 - M1.5 | -0.001 [-0.004 to 0.001] | -0.001 [-0.005 to 0.002]
  IFNg+ - CD4+ - Gag CE 7 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD4+ - Gag CE 7 - M6.5 | 0.001 [-0.001 to 0.003] | -0.003 [-0.005 to 0.001]
  IFNg+ - CD4+ - Gag p15 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag p15 - M1.5 | -0.002 [-0.002 to 0.001] | 0.028 [0.011 to 0.052]
  IFNg+ - CD4+ - Gag p15 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p15 - M6.5 | 0.013 [0.005 to 0.023] | 0.026 [0.009 to 0.079]
  IFNg+ - CD4+ - Gag p17 - M1.5: number analyzed (Participants) | 9 | 21
  IFNg+ - CD4+ - Gag p17 - M1.5 | 0 [-0.004 to 0.003] | 0.07 [0.048 to 0.098]
  IFNg+ - CD4+ - Gag p17 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p17 - M6.5 | 0.03 [0.016 to 0.062] | 0.066 [0.032 to 0.116]
  IFNg+ - CD4+ - Gag p24 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD4+ - Gag p24 - M1.5 | 0.055 [0.03 to 0.061] | 0.054 [0.04 to 0.08]
  IFNg+ - CD4+ - Gag p24 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD4+ - Gag p24 - M6.5 | 0.08 [0.051 to 0.119] | 0.053 [0.035 to 0.098]
  IFNg+ - CD8+ - Gag CE 1 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 1 - M1.5 | 0 [0 to 0.011] | 0 [-0.003 to 0.005]
  IFNg+ - CD8+ - Gag CE 1 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 1 - M6.5 | -0.002 [-0.003 to 0.007] | -0.001 [-0.003 to 0]
  IFNg+ - CD8+ - Gag CE 2 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 2 - M1.5 | 0 [0 to 0.004] | 0 [-0.003 to 0.008]
  IFNg+ - CD8+ - Gag CE 2 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD8+ - Gag CE 2 - M6.5 | -0.003 [-0.004 to 0.004] | 0 [-0.003 to 0.004]
  IFNg+ - CD8+ - Gag CE 3 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 3 - M1.5 | 0 [-0.002 to 0.007] | 0 [-0.004 to 0.006]
  IFNg+ - CD8+ - Gag CE 3 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 3 - M6.5 | 0 [-0.005 to 0.002] | 0 [-0.002 to 0.003]
  IFNg+ - CD8+ - Gag CE 4 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 4 - M1.5 | 0 [-0.003 to 0.012] | 0 [-0.002 to 0.012]
  IFNg+ - CD8+ - Gag CE 4 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 4 - M6.5 | 0 [-0.003 to 0.005] | 0 [-0.001 to 0.002]
  IFNg+ - CD8+ - Gag CE 5 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 5 - M1.5 | 0 [-0.004 to 0] | 0 [-0.002 to 0.007]
  IFNg+ - CD8+ - Gag CE 5 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 5 - M6.5 | 0 [-0.005 to 0.001] | 0.002 [-0.003 to 0.008]
  IFNg+ - CD8+ - Gag CE 6 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 6 - M1.5 | 0 [-0.004 to 0.005] | 0 [-0.003 to 0.004]
  IFNg+ - CD8+ - Gag CE 6 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag CE 6 - M6.5 | 0.001 [-0.004 to 0.008] | 0 [-0.002 to 0.002]
  IFNg+ - CD8+ - Gag CE 7 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag CE 7 - M1.5 | -0.002 [-0.003 to 0.001] | 0 [-0.002 to 0.005]
  IFNg+ - CD8+ - Gag CE 7 - M6.5: number analyzed (Participants) | 19 | 22
  IFNg+ - CD8+ - Gag CE 7 - M6.5 | -0.003 [-0.007 to 0] | 0 [-0.003 to 0.003]
  IFNg+ - CD8+ - Gag p15 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag p15 - M1.5 | 0 [-0.004 to 0.008] | 0 [-0.002 to 0.012]
  IFNg+ - CD8+ - Gag p15 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p15 - M6.5 | -0.001 [-0.005 to 0.003] | 0.002 [-0.002 to 0.016]
  IFNg+ - CD8+ - Gag p17 - M1.5: number analyzed (Participants) | 9 | 21
  IFNg+ - CD8+ - Gag p17 - M1.5 | 0 [-0.006 to 0.004] | 0.007 [0.001 to 0.022]
  IFNg+ - CD8+ - Gag p17 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p17 - M6.5 | 0 [-0.006 to 0.005] | 0.007 [0.002 to 0.022]
  IFNg+ - CD8+ - Gag p24 - M1.5: number analyzed (Participants) | 9 | 22
  IFNg+ - CD8+ - Gag p24 - M1.5 | 0.007 [0.006 to 0.018] | 0.01 [0 to 0.058]
  IFNg+ - CD8+ - Gag p24 - M6.5: number analyzed (Participants) | 20 | 22
  IFNg+ - CD8+ - Gag p24 - M6.5 | 0.005 [-0.001 to 0.061] | 0.016 [0.001 to 0.109]

19. Secondary Outcome: Binding Antibody IgG Responses Rate by the HIV-1 Binding Antibody Multiplex Assay (BAMA) by Treatment Arm [Time Frame: M6.5]
Description: The frequency of IgG binding antibody responses were measured by the HIV-1 binding antibody multiplex assay (BAMA).Samples from post-enrollment visits were declared to have positive responses if they met three conditions: (1) the MFI minus blank (MFI*) values were ≥ antigen-specific cutoff at the 1:50 dilution level (based on the 95th percentile of baseline samples as calculated by SAS PROC UNIVARIATE default method, and at least 100 MFI minus blank), (2) the MFI minus blank values were greater than 3 times the baseline (day 0) MFI minus blank values, and (3) the MFI values were greater than 3 times the baseline MFI values.
Time Frame: M6.5
Population: Immunogenicity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 + Group 4: Control 2
Number analyzed (Participants) | 22 | 20 | 4
Participants | 20 | 16 | 0

20. Secondary Outcome: Binding Antibody IgG Responses Magnitudes by the HIV-1 Binding Antibody Multiplex Assay (BAMA) by Treatment Arm [Time Frame: M6.5]
Description: The magnitude of IgG binding antibody responses were measured by the HIV-1 binding antibody multiplex assay (BAMA). Serum HIV-1-specific IgG antibody responses are measured at the 1:50 dilution against the p24gag antigen on all available samples .The a background-subtracted mean fluorescent intensity (MFI) at the 1:50 dilution were used to summarize the magnitudes at a given time-point. MFI will be used to determine the positivity of samples. Samples from post-enrollment visits are declared to have positive responses if they meet three conditions: (1) the MFI* values are greater than the antigen-specific cutoff (based on the 95th percentile of the baseline visit serum samples and at least 100 MFI), (2) the MFI* values are greater than 3 times the baseline (day 0) MFI* values, and (3) the MFI values are greater than 3 times the baseline MFI values. The values in Groups 1 and 2 are correct as currently reported.
Time Frame: M6.5
Population: Immunogenicity Population
Measure: Median (Inter-Quartile Range); unit: adjusted Mean fluorescent intensity (MFI
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 + Group 4: Control 2
Number analyzed (Participants) | 22 | 20 | 4
adjusted Mean fluorescent intensity (MFI | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1042.1 [700.4 to 1470.9]

ADVERSE EVENTS:
Time Frame: Measured through Month 12
Description: Number of Participants Reporting Adverse Events (AEs)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Control 1 | Group 4: Control 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 16/25 | 17/25 | 2/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=25) | Group 2: Vaccine (N=25) | Group 3: Control 1 (N=3) | Group 4: Control 2 (N=3)
Any Event in SOC (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 2 (2) | 1 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (General disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication of device removal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 6 (9) | 8 (11) | 1 (1) | 1 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 4 (6) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 2 (4) | 3 (4) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 4 (8) | 5 (6) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 4 (6) | 2 (2) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premenstrual dysphoric disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03181789/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03181789/SAP_001.pdf